CLINICAL TRIAL: NCT04029389
Title: Ultrasound-Guided Tibial Nerve Block vs. Local Corticosteroid Injection: A Randomized Controlled Study for Recalcitrant Plantar Fasciitis
Brief Title: Ultrasound-Guided Tibial Nerve Block vs. Local Corticosteroid Injection in Recalcitrant Plantar Fasciitis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH8
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Plantar Fascitis; Tibial Nerve; Injections; Ultrasonography
Keywords: Plantar Fascitis; Tibial Nerve; Injections; Ultrasonography
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recalcitrant Plantar Fasciitis/Conservational (Experimental): After ESWT therapy patients suffer from extreme pain will recieve only conservational therapy (26 patients)
  Interventions: Other: Conservational therapy
- Recalcitrant Plantar Fasciitis/Local (Experimental): After ESWT therapy patients suffer from extreme pain will receive local steroid injections
  Interventions: Device: Injection
- Recalcitrant Plantar Fasciitis/Tibial nerve (Experimental): After ESWT therapy patients suffer from extreme pain will receive tibial nerve block
  Interventions: Device: Tibial nerve block

INTERVENTIONS:
Device: Injection — Local corticosteroid injection
  Arms: Recalcitrant Plantar Fasciitis/Local
Device: Tibial nerve block — Tibial nerve block
  Arms: Recalcitrant Plantar Fasciitis/Tibial nerve
Other: Conservational therapy — Only exercise and foot insoles
  Arms: Recalcitrant Plantar Fasciitis/Conservational

SUMMARY:
A randomized controlled study to search for the efficiency of tibial nerve block vs local corticosteroid injection of the plantar fascia.

DETAILED DESCRIPTION:
Three groups will be formed. After ESWT therapy, if the patients still suffer from pain (> 5 points, visual analog scale(0-10points), participants will be included in the study. One group will receive conversational therapy. Second group will be treated with local corticosteroid injection. And third group will be treated with tibial nerve block. Before-treatment, after one week, after six weeks and after 3 months evaluation of the patients will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Recalcitrant plantar Fasciitis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
VAS-Pain | Three months
  A scale on 0-10 points. 0 points indicate no pain, and 10 points show worst pain ever

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yalçınkaya, Study Director — Gaziosmanpasa Taksim Training and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Training and Research Hospital, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No